CLINICAL TRIAL: NCT01368315
Title: CT 327 in the "Atopy Patch Test" Model
Acronym: CT327 AD01-09
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Creabilis SA (Industry)
Responsible Party: Dr. Eduard Vidovic, Chief Medical Officer, Creabilis
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CT 327 AD 01-09
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CT327 (Experimental): Cream
  Interventions: Drug: CT327 application
- Placebo (Placebo Comparator): Cream (Vehicle only)
  Interventions: Drug: Placebo
- Active comparator (Active Comparator): Cream
  Interventions: Drug: Active comparator
- No intervention (No Intervention)
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: CT327 application — Topical administration of 0.5 grams cream administered twice daily for ten days to one out of four test fields marked on the patient's back.
  Arms: CT327
Drug: Placebo — Topical administration of 0.5 grams cream administered twice daily for ten days to one out of four test fields marked on the patient's back.
  Arms: Placebo
Drug: Active comparator — Topical administration of an active comparator administered twice daily for ten days to one out of four test fields marked on the patient's back.
  Arms: Active comparator
Drug: No intervention — No intervention to one out of four test fields marked on the patient's back.
  Arms: No intervention

SUMMARY:
A Randomized, Double-Blind, Phase I, Single-Center Study on the Efficacy and Safety of CT 327 in the Atopy Patch Test model.

DETAILED DESCRIPTION:
The study population will include subjects with atopic dermatitis (AD) and a positive atopy patch test (APT) test at study screening. Positive responders to the APT test will enter into a treatment period of ten days during which all subjects will have three test compounds (CT 327, Placebo or an active comparator) administered twice daily to three test fields marked on patient's back. A fourth test field will act as untreated control. A challenge with the relevant aeroallergen to which the subject is responding most strongly, as assessed at screening, will take place on Day 10. Readings of APT scores will be performed at 48 and 72 hrs after the challenge and the subjects will have a end-of-study visit 2 weeks later. Local and systemic tolerance of CT327 will be assessed during the study, in addition to its potential absorption into the systemic circulation. The effects of CT327 on modulating the immune response to aeroallergens and on the expression of immunological and inflammatory markers on biopsies of the treated areas will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 66 years of age
* Able to give informed consent
* Diagnosis of atopic dermatitis and a positive atopy patch test to at least one of the following(Dermaphagoides pteronyssinus, cat dander, grass or birch pollen)

Exclusion Criteria:

* Have concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug
* Have a positive response to petrolatum
* Be immune-compromised
* Have any clinically significant abnormal clinical laboratory test results at Screening
* Have a history of malignancy except basal cell carcinoma of the skin.
* Have an active intercurrent infection
* Have applied any topical medication (including corticosteroid, calcineurin inhibitor, topical H1 and H2 antihistamines, topical antimicrobials, other medicated topical agents) or herbal preparation to the area selected for treatment within 14 days prior to study entry.
* Have received antibiotic treatment within 1 week prior to study entry
* Within 4 weeks prior to study entry, have received systemic treatment for atopic dermatitis (including systemic corticosteroids, nonsteroidals, immunosuppressants, or immunomodulating drugs, or treatment with light).
* Have received any investigational drug or been part of any clinical study within the last three months before study entry.
* Have a history of hypersensitivity or allergic reactions to any ingredient in the CT 327 formulation or to the selected active comparator or to polyethyleneglycol.
* If female, are pregnant or lactating, or intend to become pregnant during the study period
* If female, and of child-bearing potential, not taking adequate contraception to avoid pregnancy during and three months after the study.
* History of drug, alcohol or other substance abuse or other factors limiting the ability to cooperate and to comply with the study protocol

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Result of the Atopy Patch Test (APT): measurement of the eczematous skin reaction (score) after challenge with the appropriate aeroallergen, using European Task Force on Atopic Dermatitis criteria | 13 days

SECONDARY OUTCOMES:
Local and systemic tolerance of CT 327 | 7 weeks
Plasma CT327 levels | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Med. Johannes Ring, Principal Investigator — Klinik und Poliklinik für Dermatologie und Allergologie Am Biederstein, Technische Universität München, Munich, Germany
Locations (1):
- Klinik und Poliklinik für Dermatologie und Allergologie Am Biederstein Technische Universität München, Munich, Germany